CLINICAL TRIAL: NCT06784856
Title: The Effects of Augmented Reality Facilitated Education in Promoting PICC Care Knowledge, Clinical Reasoning and Learning Engagement Among Nurses
Brief Title: Effects of AR-Based Education on PICC Care Knowledge, Clinical Reasoning, and Learning Engagement in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Principal Investigator, tygh backup, Taoyuan General Hospital, Taoyuan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TYGH112093
Record Dates: First submitted 2024-12-17; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Nursing Education
Keywords: PICC care AR teaching Clinical reasoning Learning engagement Nursing education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Introduction to Updated CVAD-PICC Guidelines and Clinical Applications
  PICC Catheter Care Management of Common PICC-Related Complications Utilization of "Augmented Reality-Assisted Teaching - PICC AR Exploration APP" Interactive Online Gaming: Participants engage directly with a scenario-based game focused on PICC care, progressing through challenges within the game.
  Interventions: Other: PICC AR APP
- Control Group (Placebo Comparator): Classroom Teaching and Case Sharing Introduction to Updated CVAD-PICC Guidelines and Clinical Applications
  PICC Catheter Care Management of Common PICC-Related Complications Case Sharing on PICC Complication Management: Researchers
  Interventions: Other: Classroom Teaching and Case Sharing

INTERVENTIONS:
Other: PICC AR APP — This study utilized Vuforia software and Unity 2022 LTS as the primary development platforms to create an AR-Enhanced and Game-Assisted Teaching curriculum. The designed "PICC AR Exploration APP" was developed for both iOS and Android platforms. The PICC-related content was based on the 8th Edition of the Infusion Therapy Standards of Practice published by the Infusion Nurses Society (INS) in 2021 and the 2022 Clinical Guidelines for Vascular Access Devices.
  The required items for PICC care procedures were photographed and used to create 3D object elements and animations for developing AR scenarios and interactive gaming elements. The design and content of the "PICC AR Exploration APP" are described as follows:
  Game Design Concept:
  The "PICC AR Exploration APP" includes a learning unit system and a quiz unit system:
  Learning Unit System Content:
  Topic 1: Updates to guidelines and an introduction to clinical applications. Topic 2: PICC catheter care, dressing change steps, and techni
  Other Names: PICC AR Exploration APP
  Arms: Experimental Group
Other: Classroom Teaching and Case Sharing — Introduction to Updated CVAD-PICC Guidelines and Clinical Applications
  PICC Catheter Care Management of Common PICC-Related Complications Case Sharing on PICC Complication Management: Researchers
  Arms: Control Group

SUMMARY:
The peripherally inserted central catheter (PICC) is the preferred venous access route for patients undergoing medium- to long-term infusion therapy. PICC insertion is a common clinical nursing procedure for intravenous infusion and drug administration. However, due to its complexity and associated risks, it is crucial to assess the needs of clinical nursing staff in PICC care and to develop appropriate educational training programs. This study aims to explore the development of a novel online "Augmented Reality (AR) Scenario-Based Gamification-Assisted Teaching" intervention to enhance nurses' competence in PICC care, improving patient care quality and treatment outcomes.

This study investigates the effectiveness of AR scenario-based gamification in improving nursing staff's cognitive knowledge, clinical reasoning skills, and learning engagement in PICC care. The study employs a block randomization trial design, involving nurses from a regional hospital in northern Taiwan. The educational intervention includes classroom instruction on PICC clinical care and complication management, combined with the "PICC AR Exploration APP," which leverages interactive gaming elements within a digital learning platform.

Through scenario-based gamified teaching, learners address situational problems and select appropriate interventions, enhancing knowledge and clinical reasoning skills. The teaching program offers benefits such as flexibility for repeated practice, cost efficiency, and high portability, making it a promising approach for PICC care training and the prevention and management of catheter-related complications.

DETAILED DESCRIPTION:
Background:

With advancements in medical technology and an aging population, peripherally inserted central catheters (PICC) have become a key method for long-term intravenous therapy. As clinical demand for PICC increases, nursing staff must have strong knowledge and clinical reasoning skills to reduce catheter-related complications. However, traditional PICC training is limited by time, space, and a lack of situational diversity, making it less effective for clinical education. Augmented Reality (AR) has been introduced into medical education to provide interactive learning environments that enhance nursing skills and clinical judgment. The "PICC AR Exploration" app provides continuous training for clinical staff, effectively improving their PICC care knowledge and clinical reasoning.

Purpose:

The purpose of this study is to evaluate the effectiveness of the "PICC AR Exploration" app in enhancing nurses' knowledge of PICC care and their clinical reasoning skills.

Method:

This study adopted a block randomization design, recruiting clinical nurses from a regional teaching hospital in northern Taiwan. The experimental group received classroom teaching combined with the "PICC AR Exploration" app, while the control group received classroom teaching and case sharing. Study tools included a PICC care knowledge scale, a clinical reasoning scale, and a learning engagement scale, with assessments conducted before the intervention, after the intervention, and six weeks post-intervention.

Expected Outcome:

The study aims to determine the effectiveness of AR-assisted teaching in enhancing nurses' PICC care knowledge, clinical reasoning skills, and engagement in learning, contributing to improved patient care quality and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

Licensed Clinical Nurses Participants must hold a valid nursing license and be clinical nursing staff. Willingness to Participate Participants must be willing to participate and provide signed informed consent.

Exclusion Criteria :

Incomplete Course Participation Participants who do not complete the full course will be excluded. Nurses Not Involved in PICC Care

Nurses from units that do not perform PICC care, such as:

Traditional Chinese medicine nurses. Delivery room nurses. Pediatric nurses. Anesthesia nurses. Post-anesthesia care unit (PACU) nurses. Operating room nurses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2024-08-03 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
PICC care Knowledge scale、Clinical Reasoning Scale | 6months
  Primary Outcome Measures:
  PICC Care Knowledge Scale Description: This scale measures participants' knowledge of PICC care. Time Frame: Baseline, immediately post-intervention, 6 weeks post-intervention. Clinical Reasoning Scale Description: This scale evaluates participants' clinical reasoning skills related to PICC care.
  Time Frame: Baseline, immediately post-intervention, 6 weeks post-intervention. Learning Engagement Scale Description: Measures participants' engagement levels during the learning process.
  Time Frame: Immediately post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No